CLINICAL TRIAL: NCT01913210
Title: Effect of Ginseng on Blood Pressure: A Systematic Review and Meta-Analysis of Controlled Trials
Brief Title: Effect of Ginseng on Blood Pressure
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Vladimir Vuksan, Principal Investigator, Unity Health Toronto
Other Study IDs: MetaBPG
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Asian ginseng

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Ginseng

SUMMARY:
To determine the effect of ginseng on blood pressure control.

DETAILED DESCRIPTION:
The effect of ginseng on blood pressure control is controversial, originating from an early 1970s observational study, suggesting that ginseng may adversely effect blood pressure. Despite these early findings, extensive research has since suggested that ginseng may have a positive effect on blood pressure. The current study will help clarify present uncertainty on the effect of ginseng on blood pressure control.

This systematic review and meta-analysis will follow The Cochrane Handbook for Systematic Reviews of Interventions. MEDLINE, EMBASE, CINAHL and The Cochrane Central Register of Controlled Trials will be searched using appropriate search terms. Intervention trials that investigate the effect of ginseng on blood pressure in humans will be included.

ELIGIBILITY:
Inclusion Criteria:

* clinical trials in humans
* randomized treatment allocation
* ≥ 1 month
* suitable control
* viable endpoint data

Exclusion Criteria:

* non-human studies
* non-randomized treatment allocation
* < 1 month
* lack of a suitable control
* no viable endpoint data
* trials where ginseng is part of a multi-herbal treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hypertensive Healthy
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 1 month

SECONDARY OUTCOMES:
Diastolic Blood Pressure | 1 month
Mean Arterial Pressure | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Unity Health Toronto; John Sievenpiper, MD, PhD, Principal Investigator — Unity Health Toronto; Allison Komishon, MSc(c), Study Director — Unity Health Toronto
Locations (1):
- The Toronto 3D Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, Toronto, Ontario, Canada